CLINICAL TRIAL: NCT03784365
Title: Randomized Control Study Comparing Single-Versus Multiple-dose Antimicrobial Prophylaxis for Peroral Endoscopic Myotomy in Achalasia
Brief Title: Single-Versus Multiple-dose Antimicrobial Prophylaxis for Peroral Endoscopic Myotomy in Achalasia
Acronym: SMAPP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Consultant Gastroenterologist, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMAPP-01
Record Dates: First submitted 2018-12-20; First posted 2018-12-21 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Achalasia Cardia
Keywords: oesophageal aperistalsis
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First group (Active Comparator): This group will receive an intravenous antibiotic for three days. The first dose will be given within half hour before the POEM procedure.
  Interventions: Drug: One dose of Cefo-perazone Sulbactum
- Second group (Experimental): This group will receive only one dose of intravenous antibiotic within half hour before the POEM procedure
  Interventions: Drug: One dose of Cefo-perazone Sulbactum

INTERVENTIONS:
Drug: One dose of Cefo-perazone Sulbactum — Antibiotic
  Other Names: Multiple doses of Cefo-perazone Sulbactum

SUMMARY:
Achalasia cardia is a primary oesophageal motility disorder of unknown etiology. Recently, peroral endoscopic myotomy (POEM) has gained widespread acceptance as an effective treatment modality for achalasia.

Major adverse events are uncommon with POEM. Since the operator works close to mediastinum during the POEM procedure, there is a potential for infectious complications. Therefore, intravenous antibiotics are universally used to prevent infection-related adverse events. There is no fixed protocol or duration of antibiotics for the same.

DETAILED DESCRIPTION:
POEM is a novel minimally invasive treatment for achalasia, which emerged as an offshoot of natural orifice transluminal endoscopic surgery (NOTES). Major adverse events during POEM are rare and therefore, the procedure is considered safe.

Bacteremia can occur after endoscopic procedures like esophageal dilation, sclerotherapy of varices, and instrumentation of obstructed bile ducts. Bacteremia has been advocated as a surrogate marker for risk of infection-related complications. In POEM procedure, the endoscopist works in close proximity to mediastinum and peritoneal cavity. Therefore, the potential for infection-related complications is high. However, despite of different antibiotic protocols at different centers, the reported incidence of infection-related complications is very low. At present, prophylactic antibiotics are universally initiated before starting the POEM procedure and continued for a variable duration after POEM ranging from 1 day to 7 days.

Data from surgical studies indicate that prolonged administration of antibiotics for longer than 24 hours may not be beneficial. Prolonged use of antibiotics not only increases the costs and exposure to drug toxicity directly but also may be associated with an increased risk of acquired antibiotic resistance as well as infection with Clostridium difficile.

With this background, we planned a study to evaluate the difference in the infectious complications between short vs long duration antibiotic in patients with achalasia undergoing POEM.

ELIGIBILITY:
Inclusion Criteria:

* All the patient(aged 18-65) who underwent POEM for achalasia cardia.

Exclusion Criteria:

* Unwillingness to give written informed consent

  * Patients with multiple co morbidities.
  * Immunocompromised patients /on steroid therapy.
  * Patients with indications for antibiotic prophylaxis (infective endocarditis).
  * Patients who have received antibiotics in the last 1 week .
  * Patients who have possible signs of infection during preparation for POEM

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Infectious complications associated with POEM | 1 month
  The primary outcome of the study is to estimate the difference in the incidence of infectious complications in the two groups

SECONDARY OUTCOMES:
Incidence of positive blood cultures | 72 hours
  The main secondary outcome is difference in the incidence of positive blood cultures between the two groups
Comparison of serum Procalcitonin between the two groups | 72 hours
  Difference in the mean serum procalcitonin values between both the groups
Comparison of inflammatory markers (CRP) between the two groups | 72 hours
  Both the groups will be compared for mean blood C-reactive protein (CRP)
Comparison of erythrocyte sedimentation rate (ESR) between the two groups | 72 hours
  Both the groups will be compared for mean ESR at 1-hour
Adverse events associated with administration of intravenous antibiotics | 1-month
  Both the groups will be compared for the incidence of complications associated with the use of intravenous antibiotics

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Ramchandani, Principal Investigator — Asian Institute of Gastroenterology, Hyderabad, India
Locations (1):
- Dr.Mohan Ramchandani, Hyderabad, RED ROSE Restaurant, India

REFERENCES:
- [Derived] Nabi Z, Bhaware B, Ramchandani M, Basha J, Inavolu P, Kotla R, Goud R, Darisetty S, Reddy DN. Single-Versus Multiple-Dose Antimicrobial Prophylaxis in Peroral Endoscopic Myotomy: A Randomized Controlled Study (SMAPP Trial). Dysphagia. 2023 Dec;38(6):1581-1588. doi: 10.1007/s00455-023-10585-y. Epub 2023 May 4. PMID 37142733